CLINICAL TRIAL: NCT01658956
Title: A Phase II Randomized Study to Verify the Papaldo's Hypothesis : the Effectiveness of a Reduced Dosing of G-CSF in Chemotherapy-treated Patients With a Low to Moderate Risk of Febrile Neutropenia
Brief Title: Effectiveness of Reduced GCSF Dosing in Patients With a Low to Moderate Risk of Febrile Neutropenia
Acronym: PAPALDO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Institut Jules Bordet
Record Dates: First submitted 2012-07-27; First posted 2012-08-07 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
Keywords: GCSF; Chemotherapy; Breast cancer; Prophylaxis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous GCSF 5 µg/kg days 8 and 12 (Experimental): Prophylactic administration of GCSF on days 8 and 12 following chemotherapy
  Interventions: Drug: GCSF administration on days 8 and 12 after chemotherapy
- No intervention (No Intervention)

INTERVENTIONS:
Drug: GCSF administration on days 8 and 12 after chemotherapy
  Arms: Subcutaneous GCSF 5 µg/kg days 8 and 12

SUMMARY:
The study aims to confirm that a reduced dosage of GCSF is effective in preventing febrile neutropenia among patients with breast cancer, treated with chemotherapy and presenting with a low to moderate risk of developing febrile neutropenia.

ELIGIBILITY:
Inclusion Criteria:

Breast cancer Chemotherapy administration (new line) Chemotherapy type : FEC, EC, AC, docetaxel containing regimen Chemotherapy setting : adjuvant or neoadjuvant

Exclusion Criteria:

Eligibility to receive reimbursed GCSF

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a febrile neutropenic episode defined as fever (>=38.5°C once or >=38°C twice within 12 hours interval) and neutropenia (ANC < 0.5 IU) | At the beginning of 2nd chemotherapy cycle, no more than 30 days after randomization

SECONDARY OUTCOMES:
Need for unplanned hospitalization | At the beginning of second chemotherapy cycle, no more than 30 days after randomization
  Unplanned hospitalization is defined as the need to admit a patient outside of the schedule that was planned for chemotherapy administration
Complicated febrile neutropenic episode | At the beginning of the second chemotherapy cycle, no more than 30 days after randomization
  A complicated febrile neutropenic episode is defined as a febrile neutropenic episode (see above) that does not resolve without the occurrence of serious medical complication as defined in Klasterky J et al; JCO 2000 : 3038-3051
Mortality any cause | 30 days from randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium